CLINICAL TRIAL: NCT07130539
Title: Mediterranean-DASH Intervention for Neurodegenerative Delay and High-Intensity Interval Training to Improve Blood Pressure and Other Cardiovascular Disease Risk Factors in Adults With Hypertension and Overweight/Obesity
Brief Title: Mediterranean-DASH Intervention for Neurodegenerative Delay and High-Intensity Interval Training in Adults With Hypertension
Acronym: MIND HIIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Wesley Tucker, Associate Professor of Nutrition, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY2025-184
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hypertension (HTN); Obesity &Amp; Overweight; Sedentary
Keywords: Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND); High-Intensity Interval Training (HIIT); Hypertension; Sleep; Nocturnal Blood Pressure; Ambulatory Blood Pressure Monitoring; Lifestyle Intervention; Overweight/Obesity; Cardiovascular Disease; Inflammation; Extra Virgin Olive Oil; Nuts
MeSH Terms: conditions — Hypertension; Obesity; Overweight; Sedentary Behavior; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Intervention Model Description: Pilot/Feasibility Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MIND Diet + High-Intensity Interval Training (HIIT) (Experimental): 4 week intervention consisting of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet and High-Intensity Interval Training (HIIT) Exercise
  Interventions: Other: MIND HIIT

INTERVENTIONS:
Other: MIND HIIT — 4 week intervention consisting of the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) Diet in combination with 3 days per week of High-Intensity Interval Training (HIIT) exercise

SUMMARY:
This pilot study examines whether a 4-week diet and exercise intervention can improve blood pressure, heart health, and sleep in physically inactive individuals with high blood pressure and overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 74 years old
* BMI 25 - 39.9 kg/m2 (for measured BMI)
* Clinically diagnosed hypertension (physical medical record showing diagnosis of hypertension) with or without current medication use (SPB < 160 mm Hg, DBP < 100 mm Hg)
* Physically inactive < 7,500 steps per day (measured on Fitbit over 1-week)
* No current injury, illness, or joint issue that prevents participation in exercise
* Able to read and speak English
* Willingness to participate and give informed written consent
* Willingness to share medical record indicating diagnosis of HTN and current medication use

Exclusion Criteria:

* Pregnant, breastfeeding, lactating
* Current smoker
* Food allergy or lactose intolerance
* Height > 6 foot 6 inches (78 inches)
* Blood pressure ≥ 160/100 mm Hg (Contraindication to exercise testing)
* History of diagnosed cardiovascular diseases including heart attack, stroke, irregular heartbeat such as atrial fibrillation, coronary artery or peripheral artery disease, or heart failure
* History of liver, kidney, or metabolic disease (including type I or II diabetes)
* History of cancer
* Diagnosed moderate to severe obstructive sleep apnea, CPAP use, insomnia, h/o other sleep disorder
* Night shift and/or rotating shift worker (current or in the past 2 years)
* Current use of sleep medications or sleep aids
* Excessive alcohol intake - ≥ 8 drinks per week in women, ≥ 15 drinks per week in men
* History of gastric bypass or other weight loss surgery
* Current use of metformin, insulin, dietary supplements or drugs for glycemic control or weight loss
* Weight stable for the last 2 months (< 5 pounds body weight change)
* Currently following a special diet for weight loss (Keto, Atkins, Intermittent Fasting)
* A "yes" response to any questions on the PAR-Q (excluding Question 6 on use of BP medications)
* Exercise training (≥ 2 days per week structured aerobic and resistance training at gym)
* Prior hospitalization for COVID-19
* Any medications or supplements that may alter study outcomes as determined by study PI

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-08-23 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT in adults with HTN and overweight/obesity. | From baseline to end of treatment at 4 weeks
  Adherence to the lifestyle intervention will be determined by ≥ 75% supervised exercise training visits completed and ≥ 75% dietary compliance.

SECONDARY OUTCOMES:
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to lower blood pressure in adults with HTN and overweight/obesity. | Baseline and end of intervention at 4 weeks
  Clinic-based blood pressure will be measured in triplicate at each testing visit using a Welch Allyn Automated Blood Pressure Unit and 24-hour blood pressure will also be measured using SunTech Oscar 2 Ambulatory Blood Pressure Monitors
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to improve nocturnal blood pressure in adults with HTN and overweight/obesity. | At baseline and at the end of the 4 week intervention
  Nocturnal blood pressure will be measured using SunTech Oscar 2 Ambulatory Blood Pressure Monitors
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to improve cardiorespiratory fitness in adults with HTN and overweight/obesity. | Baseline and end of intervention at 4 weeks
  Cardiorespiratory fitness will be assessed via maximal oxygen uptake (VO2max) on a cycle ergometer
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to improve cardiometabolic blood biomarkers in adults with HTN and overweight/obesity. | At baseline and end of the intervention at 4 weeks
  Fasting blood will be drawn, processed, and analyzed for glucose, insulin, lipids, and inflammatory markers.
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to lower visceral fat in adults with HTN and overweight/obesity. | Baseline and end of intervention at 4 weeks
  Visceral fat will be measured via dual-energy x-ray absorptiometry (DEXA)
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to improve quality of life in adults with HTN and overweight/obesity. | Baseline and at the end of the intervention at 4 weeks
  Health-related quality of life will be measured with the 36-item Short-Form Health Survey (SF-36)

OTHER OUTCOMES:
To evaluate the efficacy of a 4-week novel lifestyle intervention consisting of a MIND diet and HIIT to improve sleep quality in adults with HTN and overweight/obesity. | At baseline and at the end of the 4 week intervention
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) and Fitbit Inspire 3 trackers.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's University Houston Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, ICF
Time Frame: July 2026 to July 2028
Access Criteria: Email study PI

DOCUMENTS (2):
  • Study Protocol (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT07130539/Prot_000.pdf
  • Informed Consent Form (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT07130539/ICF_001.pdf